CLINICAL TRIAL: NCT05198414
Title: SER+ Against COVID-19 - Interventions to Strengthen the Resilience of Organizations and Professionals of the Public Health System in Ecuador.
Brief Title: SER+ Against COVID-19 - Interventions to Strengthen the Resilience of HCWs in Ecuador
Status: Completed | Type: Observational
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Universidad Catolica Santiago de Guayaquil (Other); Hospital General del Norte de Guayaquil IESS Los Ceibos (Unknown)
Responsible Party: Principal Investigator, José Joaquín Mira, Professor, Universidad Miguel Hernandez de Elche
Other Study IDs: UMHODS22
Record Dates: First submitted 2022-01-17; First posted 2022-01-20 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Occupational Stress; Stress, Physiological
Keywords: Healthcare workers; Qualitative study; COVID-19; Quality of care; Occupational Stress; Stress, Physiological
MeSH Terms: conditions — Occupational Stress; COVID-19 | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: Healthcare workers at the first line and healthcare directives.
  Interventions: Other: Focus group

INTERVENTIONS:
Other: Focus group — Qualitative research methodology with healthcare workers

SUMMARY:
The SARS-CoV-2 pandemic has particularly impacted Ecuador. By May 31, 2021, 426,000 cases (10% of health professionals) and 20,572 deaths. Care procedures, organization and priorities have been altered, if not broken. The quality and safety of COVID19 and non-COVID19 patients have been compromised. Compassion fatigue, post-traumatic stress and moral damage reactions have been observed among healthcare professionals, considered second victims of SARS-CoV-2. Without professionals who feel supported and morally strong, care will be compromised, leading to greater uncertainty and insecurity in the care of COVID19 and non-COVID19 patients. In coordination with local authorities, this project seeks to strengthen the resilience of public institutions and healthcare professionals to implement. In coordination with local authorities, this project seeks to strengthen the resilience of public institutions and health professionals to implement proven interventions and scale them up to the whole health system to strengthen it after the impact of the COVID19 pandemic. This proposal is aligned with Sustainable Development Goal 3, which includes different targets to ensure healthy lives and promote well-being for all ages. Health emergencies, such as the one resulting from COVID-19, pose a global risk and have shown that preparedness is vital. Improving the Quality of the National Health Services and strengthening the health system in preparedness and response to health emergencies are the main priority lines of action in this project, thus aligning with SDG target 3.8 concerning strengthening health professional morale since to save lives, countries' public health systems must be strengthened. Previous work with the local partner supports the good performance and development of this proposal, which arose from a need based on the need to This proposal arose from a need based on the lessons learned in Spain.

DETAILED DESCRIPTION:
The COVID-19 pandemic has been one of the health emergencies with the most significant impact on the world's population as a whole since records have been kept. The number of infected people (more than 234 million cases as of October 5, 2021) and deaths from this cause (4.8 million as of October 5, 2021) had exceeded any initial forecast when the WHO declared a public health emergency of international concern on January 30, 2020, and subsequently reported the COVID-19 outbreak a pandemic on March 11, 2020. In Ecuador, the situation has been equally alarming, with excess mortality of 46,470 people, which proportionally represents an increase of 57.72% compared to 2019 during 2020. As of December 6, 526,000 cases and 33,000 deaths have been confirmed.

Health organizations in Ecuador have faced this health crisis by implementing organizational and structural reforms (for example, increasing the number of beds in critical care units to the limit of possibilities and setting up convention centers for the care of COVID patients). No specific measures have been put in place to alleviate pressure and help professionals cope with compassion fatigue or acute stress experienced during the most critical moments of the pandemic. This situation was exacerbated by the scarcity of personal protective equipment, fear, and distress of health professionals as they put their lives and their family members at risk.

This study aims to draw lessons learned from these responses that have contributed to dealing with the health emergency, both at the institutional and individual level of health personnel, identifying those actions that have had a positive impact. These lessons can be used in the future in other crises and emergencies to develop measures for the protection and organization of the work of health personnel and to achieve a better response for the benefit of patients.

This perspective-shifting approach focuses on the positive things that have helped health professionals cope with the pandemic that has not been sufficiently researched previously. Most studies focus on the negatives and what has gone wrong, but it is time to look back and compile the things that have helped us have valuable tools for future public health emergencies.

Methods Mixed study that combines a first phase of qualitative research with a second phase of field study to, through a survey, capture information relevant to the objectives of the study and, finally, to develop a series of recommendations to support Ecuador's health system in the post-pandemic of COVID-19 and increase the resilience of personnel in future health emergencies.

First phase

The Focus Group technique will be used to capture experiences, experiences and measures taken to cope with the emotional consequences of the pandemic among the staff of the different health centers. We will seek to include primary care and hospital professionals from the city of Guayaquil. Group sessions will be conducted, each with between 8 and 11 participants, and the dynamics will be maintained until information saturation is reached. Recruitment will be carried out using the snowball technique among health professionals (physicians, nurses, support staff, among others). These group sessions will be complemented with a minimum of 5 and a maximum of 10 semi-structured interviews with middle managers of the organization and managers of at the level of the Integral Public Health Network (RSPI), such as the Ecuadorian Institute of Social Security, a health care referent and the North General Hospital of Guayaquil. The latter became a sentinel hospital for the care of most of the cases during this pandemic. For this reason, it has been considered ideal for conducting focus groups and surveys. The discourse will be analyzed and the ideas will be classified into categories. The information obtained will be triangulated and its consistency will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers of primary care providng care to COVID-19 patients.
* Healthcare workers of hospitals providng care to COVID-19 patients.
* Medical directors (high management) of COVID-19 hospitals.
* Administrative personnel of COVID-19 hospitals.

Exclusion criteria:

- Healthcare workers, medical directors and administrative personnel not involved in COVID19 care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health professionals of primary care, hospital, medical directors and administrative personnel of the city of Guayaquil who have been working directly with COVID patients or in facilities destined to the care of COVID patients.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Recommendations to support and increase the resilience of healthcare workers | 31/05/2022
  Recommendations to support Ecuador's health system in the COVID-19 pandemic and increase the resilience of personnel in future health emergencies.

OTHER OUTCOMES:
Categories of analysis | 01/02/2022
  Capture experiences, feelings and measures taken to cope with the emotional consequences of the pandemic among healthcare workers

CONTACTS AND LOCATIONS:
Overall Officials: Jose J Mira Solves, PhD, Principal Investigator — Universidad Miguel Hernandez
Locations (2):
- Ecuador (2):
  - Hospital General Norte "Los Ceibos", Guayaquil, Guayas
  - Universidad Católica de Santiago de Guayaquil, Guayaquil, Guayas

IPD SHARING:
Plan to Share IPD: No
As this is a qualitative study, participants' data, verbatims, and transcription of recorded focus groups can not be disclosed.

REFERENCES:
- [Background] Mira JJ, Carrillo I, Guilabert M, Mula A, Martin-Delgado J, Perez-Jover MV, Vicente MA, Fernandez C; SARS-CoV-2 Second Victim Study Group. Acute stress of the healthcare workforce during the COVID-19 pandemic evolution: a cross-sectional study in Spain. BMJ Open. 2020 Nov 6;10(11):e042555. doi: 10.1136/bmjopen-2020-042555. PMID 33158839
- [Background] Martin-Delgado J, Viteri E, Mula A, Serpa P, Pacheco G, Prada D, Campos de Andrade Lourencao D, Campos Pavan Baptista P, Ramirez G, Mira JJ. Availability of personal protective equipment and diagnostic and treatment facilities for healthcare workers involved in COVID-19 care: A cross-sectional study in Brazil, Colombia, and Ecuador. PLoS One. 2020 Nov 11;15(11):e0242185. doi: 10.1371/journal.pone.0242185. eCollection 2020. PMID 33175877
- [Result] Mira JJ, Vicente MA, Lopez-Pineda A, Carrillo I, Guilabert M, Fernandez C, Perez-Jover V, Martin Delgado J, Perez-Perez P, Cobos Vargas A, Astier-Pena MP, Martinez-Garcia OB, Marco-Gomez B, Abad Bouzan C. Preventing and Addressing the Stress Reactions of Health Care Workers Caring for Patients With COVID-19: Development of a Digital Platform (Be + Against COVID). JMIR Mhealth Uhealth. 2020 Oct 5;8(10):e21692. doi: 10.2196/21692. PMID 32936769
- [Result] Mira JJ, Cobos-Vargas A, Astier-Pena MP, Perez-Perez P, Carrillo I, Guilabert M, Perez-Jover V, Fernandez-Peris C, Vicente-Ripoll MA, Silvestre-Busto C, Lorenzo-Martinez S, Martin-Delgado J, Aibar C, Aranaz J. Addressing Acute Stress among Professionals Caring for COVID-19 Patients: Lessons Learned during the First Outbreak in Spain (March-April 2020). Int J Environ Res Public Health. 2021 Nov 16;18(22):12010. doi: 10.3390/ijerph182212010. PMID 34831767
- See also: Social Observatory of Ecuador. Deceased persons — https://www.covid19ecuador.org/fallecidos
- See also: World Health Organization (WHO). WHO Coronavirus Disease (COVID-19) Dashboard — https://covid19.who.int